CLINICAL TRIAL: NCT03634631
Title: Effects of Transcranial Focused Ultrasound on Human Primary Motor Cortex Using 7T fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1508M77355
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Ultrasound in MRI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Focused Ultrasound — Test ultrasound in 7T MRI scanner

SUMMARY:
Transcranial focused ultrasound (tFUS) is a form of neuromodulation that uses a single element transducer to produce highly focused low-intensity acoustic energy that can be used to affect cortical excitability in humans. This technology has an advantage over existing electric and electromagnetic technologies in that it has very high spatial resolution and can be focused deep to the cortical surface to target sub-cortical neural structures and circuits. Previous research has shown that tFUS can affect human tactile detection thresholds (Legon et al. 2014a) as well as functional measures of the electroencephalogram (EEG) (Legon et al. 2014a; Mueller et al. 2014a). However, EEG does not provide for detailed spatial mappings and thus the specific spatial extent of the effect of acoustic energy in the cortex is not yet understood. This is an important consideration for the advancement of tFUS as a non-surgical method of stimulation of discrete cortical circuits and small sub-cortical neural structures. Is the effect of tFUS limited to its beam maxima? Does the effect extend along the beam path? And if so, to what extent? These questions can be answered if tFUS is combined with magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Background and Significance:

MRI provides highly detailed spatial maps of cortical and sub-cortical activation. As such, delivering tFUS in the MR scanner can provide critical information on neural activation as a result of tFUS. It is unclear however, if tFUS can generate a detectable blood-oxygen level dependent (BOLD) response. Preliminary evidence in humans (Mueller et al. 2014b; Legon et al. 2015) has demonstrated mostly negative results and highly variable responses perhaps due to the transducer or acoustic intensity levels used, the pulsing strategy employed and/or poor signal to noise ratios. We know from animal work it is possible to detect a change in BOLD response from tFUS if a known signal already exists. Yoo et al. (2011) showed focused ultrasound to attenuate the BOLD signal generated by visual stimuli in visual cortex of rabbits. Thus, it is reasonable to assume that this effect is transferable to humans as the underlying brain physiology producing the BOLD signal is the same.

Here we plan to investigate the effect of tFUS on the BOLD signal in human primary motor (M1). M1 has been chosen for two fundamental reasons. 1) The use of muscle contraction to generate a BOLD signal in M1 allows for investigation tFUS on the peripheral electromyogram (EMG) and 2) spatially specific BOLD responses in the cortex can be generated depending upon the musculature used, thus allowing for precise spatial mapping of effect. The first point is of significant interest because if a detectable effect is demonstrated on peripheral musculature it provides important initial evidence that tFUS operates on cortical motor neurons and descending motor tracts similar to electric and electromagnetic stimulation thus hinting at the cellular populations and mechanisms affected by and responsible for tFUS neuromodulatory effect. The second point confirms with high precision the spatially selective effect of tFUS and if we can establish energy/effect functions from this data, this can also lead to scaling of tFUS energies to elicit specific effects such as inhibition or excitation.

Together, this knowledge will further promote tFUS for cortical stimulation and progress tFUS for subcortical stimulation in humans. This last advancement is the great potential of tFUS. Imagine a small device that can simply be attached to the head for precise stimulation anywhere in the brain in lieu of surgery. This is the ultimate goal of this research, however, before this can be considered, the detailed data from this research proposal is necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age Provide written informed consent

Exclusion Criteria:

* Evidence of a current significant medical illness or psychiatric or central or peripheral neurologic disorder History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services Personal or family history of seizure Any history of stroke/transient ischemic attack (TIA) Taking any medications that may decrease the threshold for seizure Pregnancy Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI Failure to follow laboratory or study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Primary motor cortex BOLD signal | 30 minutes
  Primary motor cortex BOLD signal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ai L, Bansal P, Mueller JK, Legon W. Effects of transcranial focused ultrasound on human primary motor cortex using 7T fMRI: a pilot study. BMC Neurosci. 2018 Sep 14;19(1):56. doi: 10.1186/s12868-018-0456-6. PMID 30217150